CLINICAL TRIAL: NCT00202423
Title: fMRI and Neurophysiological Study Protocol on Cannabinoids in Multiple Sclerosis
Brief Title: Use of Cannabinoids in Patients With Multiple Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: S. Andrea Hospital (Other)
Collaborators: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-CAN-04; CRI.FS032
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-11-29 (Estimated); Status verified 2005-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Cannabinoids; Spasticity; fMRI; TMS
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity | interventions — nabiximols

INTERVENTIONS:
Drug: Sativex

SUMMARY:
This is a 10-week, randomised, double blind, placebo-controlled, crossover trial to investigate the effect of Cannabis Based Medicine Extract (Sativex) on patterns of brain activation associated with movement in 20 MS patients suffering from lower limb spasticity. Spasticity is a common symptom in Multiple Sclerosis (MS), occurring all over the course of the disease, particularly in the progressive phase.Physiologically, spasticity and hyperreflexia habitually seen in patients with pyramidal syndrome is due to lesions of other descending pathways, such as the cortico reticulospinal pathways, which participate in voluntary movements.It is now known that an endocannabinoid system acts in humans by at least two types of cannabinoids receptors, CB1 and CB2. There is evidence to support the view that the psychoactive ingredient in cannabis, delta 9-tetrahydrocannabinol (delta 9-THC), and cannabinoids in general, can reduce muscle spasticity in people with MS. Aim of the study will be to evaluate the effect of Sativex on: (i) patterns of brain activation associated with movement (fMRI) in MS patients suffering from spasticity; (ii) changes in level of spasticity (H-reflex); (iii) changes in intracortical excitability and on synaptic intracortical network of the motor areas (double shock TMS).

DETAILED DESCRIPTION:
Baseline assessment will be followed by randomisation and dose introduction. Patients will be randomly assigned to two counterbalanced groups starting either with Sativex or with placebo as the first drug. They will be dispensed sufficient study medication for two weeks together with a diary. During the two-week treatment period all the patients will have to be reached the optimal, individualised dosage to subjectively relief spasticity.Patient will return after three weeks and they will undergo the fMRI and neurophysiological evaluations.Then patients will perform a two-week washout period and they will be requested to intake the alternative medicine. After two weeks patients will perform a second fMRI/neurophysiological study. Two weeks later, after a second washout period, a last visit will be performed to conclude the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 60 years of age (inclusive)
2. Have definite Multiple Sclerosis as per Poser Criteria
3. Have either relapsing remitting or secondary progressive course
4. Baseline EDSS score from 3.0 to 6.5 (inclusive)
5. Stable disease for at least 30 days prior to study entry
6. Be right-handed with normal right hand function
7. Female patients of child bearing potential and male patients whose partner is of child bearing potential who are willing to ensure that they or their partner use effective contraception during the study and for three months thereafter
8. If female, be neither pregnant nor breast-feeding. Confirmation that the subjects not pregnant must be established by a negative serum hCG pregnancy test at baseline.
9. No cannabinoids use (cannabis, Marinol, Nabilone) for at least three months prior to entry into the study and willing to abstain from any use of cannabis during the study
10. Significant spasticity in at least two muscle groups defined as a score of 2 or more on the Ashworth scale for each muscle group
11. Antispastic/antiepileptic treatments (dosage, frequency and route of administration) stable for at least one month prior the study entry

    -

Exclusion Criteria:

1. Have a primary progressive MS
2. Patients under disease modifying therapies prescribed in the 6 months prior the study entry
3. Patients who have participated in another research study in the past 6 months
4. Changes in antispastic/antiepileptic treatments (dosage, frequency and route of administration) within one month prior the study entry
5. Have a psychiatric disorders or cognitive impairment that preclude safe participation in the study
6. Known history of alcohol or substance abuse
7. Concurrent clinically important immunologic, pulmonary, renal, liver, active thyroid, and/or other major disease other than MS
8. Severe cardiovascular, disorders, such as ischaemic heart disease, arrhythmias, poorly controlled hypertension or severe heart failure
9. Patients suffering from acute or chronic pain
10. History of epilepsy
11. Female patient who is pregnant, lactating or planning pregnancy during the course of the study
12. Scheduled elective surgery or other procedures requiring general anaesthesia during the study
13. Patient who is terminally ill or is inappropriate for placebo medication
14. Systemic corticosteroid therapy within 4 weeks of randomization or exacerbation of MS within 30 days
15. Regular levodopa therapy within 7 days of the study entry
16. Male patient currently receiving sildenafil (Viagra) and unwilling to stop medication for the duration of the study
17. Patients who are currently taking antiarrhythmic medications
18. Known or suspected adverse reaction to cannabinoids
19. Travel outside the Italy planned during the study
20. Donation of blood during the study
21. Contraindications to MRI scans -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-07

PRIMARY OUTCOMES:
To evaluate the effect of Sativex on: a)patterns of brain activation associated with movement(fMRI); b) changes in level of spasticity (H-reflex); c)changes in intracortical excitability and on synaptic intracortical network of the motor areas(TMS).

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Inghilleri, MD, Principal Investigator — Policlinico Umberto I, University of Rome "La Sapienza"; Carlo Pozzilli, MD, Study Director — Policlinico Umberto I, University of Rome "La Sapienza"
Locations (1):
- Department of Neurology- University of Rome la Sapienza, Rome, Italy

REFERENCES:
- [Background] Pertwee RG. Cannabinoid receptor ligands: clinical and neuropharmacological considerations, relevant to future drug discovery and development. Expert Opin Investig Drugs. 2000 Jul;9(7):1553-71. doi: 10.1517/13543784.9.7.1553. PMID 11060760
- [Background] Smith PF. Cannabinoids in the treatment of pain and spasticity in multiple sclerosis. Curr Opin Investig Drugs. 2002 Jun;3(6):859-64. PMID 12137404
- [Background] Zajicek J, Fox P, Sanders H, Wright D, Vickery J, Nunn A, Thompson A; UK MS Research Group. Cannabinoids for treatment of spasticity and other symptoms related to multiple sclerosis (CAMS study): multicentre randomised placebo-controlled trial. Lancet. 2003 Nov 8;362(9395):1517-26. doi: 10.1016/S0140-6736(03)14738-1. PMID 14615106
- [Background] Baker D, Pryce G, Croxford JL, Brown P, Pertwee RG, Huffman JW, Layward L. Cannabinoids control spasticity and tremor in a multiple sclerosis model. Nature. 2000 Mar 2;404(6773):84-7. doi: 10.1038/35003583. PMID 10716447
- [Background] Wade DT, Robson P, House H, Makela P, Aram J. A preliminary controlled study to determine whether whole-plant cannabis extracts can improve intractable neurogenic symptoms. Clin Rehabil. 2003 Feb;17(1):21-9. doi: 10.1191/0269215503cr581oa. PMID 12617376
- [Background] Wade DT, Makela P, Robson P, House H, Bateman C. Do cannabis-based medicinal extracts have general or specific effects on symptoms in multiple sclerosis? A double-blind, randomized, placebo-controlled study on 160 patients. Mult Scler. 2004 Aug;10(4):434-41. doi: 10.1191/1352458504ms1082oa. PMID 15327042
- [Background] Vaney C, Heinzel-Gutenbrunner M, Jobin P, Tschopp F, Gattlen B, Hagen U, Schnelle M, Reif M. Efficacy, safety and tolerability of an orally administered cannabis extract in the treatment of spasticity in patients with multiple sclerosis: a randomized, double-blind, placebo-controlled, crossover study. Mult Scler. 2004 Aug;10(4):417-24. doi: 10.1191/1352458504ms1048oa. PMID 15327040